CLINICAL TRIAL: NCT02911870
Title: A Thorough QTc Trial Evaluating the Effect of SNAC on Cardiac Repolarisation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4247; 2015-002418-54 (EudraCT Number); U1111-1170-7054 (Other: WHO)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A, SNAC (Experimental): Single dose of 1.2mg, 2.4mg or 3.6mg increasing for each cohort of trial participants.
  Interventions: Drug: SNAC
- Part A, placebo (Placebo Comparator): Single dose at corresponding dose levels.
  Interventions: Drug: Placebo
- Part B, SNAC, Placebo, Moxifloxacin (Experimental): Subjects will receive 4 different treatments in random order. SNAC dose between 1.2-3.6 mg, Placebo in two different periods, moxifloxacin 400mg.
  Interventions: Drug: SNAC; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: SNAC — Oral administration
  Arms: Part A, SNAC; Part B, SNAC, Placebo, Moxifloxacin
Drug: Placebo — Oral administration
  Arms: Part A, placebo; Part B, SNAC, Placebo, Moxifloxacin
Drug: Moxifloxacin — Oral administration
  Arms: Part B, SNAC, Placebo, Moxifloxacin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the effect of SNAC on cardiac repolarisation in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 18.5-28.0 kg/m^2 (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs and clinical laboratory tests performed during the screening visit, as judged by the investigator
* Normal electrocardiogram (ECG) at screening or minor findings considered not clinically significant, as judged by the investigator

Exclusion Criteria:

* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per week), or subject smoking equal to or less than 5 cigarettes or the equivalent per week who is not able or willing to refrain from smoking and use of nicotine substitute products within 48 hours prior to each dosing and during the in-patient periods
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening
* Sitting blood pressure at screening (after resting for at least 5 minutes) outside the range of 90-139 mmHg for systolic or 50-89 mmHg for diastolic
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy,gastric bypass surgery)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From dosing (day 1) to follow-up (days 8-11)
  PART A
The co-primary endpoints are Fridericia heart rate corrected QT interval (QTcF) | At 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 8, and 12 hours
  PART B

SECONDARY OUTCOMES:
Maximum observed SNAC plasma concentration | From 0 to 12 hours
  PART A
Trial population-specific (accounted for individual subject levels) corrected QT interval (QTcP) | At 10, 20, 30, 40, 50 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 8 and 12 hours
  PART B
Area under the SNAC plasma concentration time curve | From 0 to 12 hours
  PART B
Maximum observed SNAC plasma concentration | From 0 to 12 hours
  PART B

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Granhall C, Baekdal TA, Breitschaft A, Sondergaard FL, Anderson TW, Thomsen M. Absence of QTc Prolongation with Sodium N-(8-[2-Hydroxybenzoyl] Amino) Caprylate (SNAC), an Absorption Enhancer Co-Formulated with the GLP-1 Analogue Semaglutide for Oral Administration. Diabetes Ther. 2021 Sep;12(9):2599-2610. doi: 10.1007/s13300-021-01106-x. Epub 2021 Jul 28. PMID 34319564